CLINICAL TRIAL: NCT03284918
Title: Effect of a Cereal Based Snack Bar With Added Plant Stanol Ester on Serum Total and Lipoprotein Lipids
Brief Title: Lipid Lowering Effect of a Cereal Based Snack Bar With Added Plant Stanol Ester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Collaborators: Oy Medfiles Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MFRA004
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Plant stanol ester (Experimental): Cereal based snack bar with added plant stanol ester (0.8 g plant stanols/bar). Two bars consumed daily as a snack, between meals, for 4 weeks (1.6 g plant stanols/d).
  Interventions: Dietary Supplement: Plant stanol ester
- Placebo (Placebo Comparator): Cereal based snack bar without plant stanol ester. Two bars consumed daily as a snack, between meals, for 4 weeks (0 g plant stanols/d).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant stanol ester
  Arms: Plant stanol ester
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the cholesterol lowering efficacy of a cereal based snack bar with added plant stanol ester when used between meals as part of a habitual diet by subjects with mild to moderate hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Serum total cholesterol 5.2-8.5 mmol/l
* Serum triglycerides < 3 mmol/l
* Signed written informed consent

Exclusion Criteria:

* Abnormal liver, kidney and thyroid function
* Use of lipid lowering medication
* Consumption of other plant sterol or plant stanol containing food products or supplements, or other foods or supplements for cholesterol lowering 1 month prior to visit 2
* History of unstable coronary artery disease (myocardial infarction, coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA) within the previous 6 months
* Diagnosed type 1 or type 2 diabetes requiring medical treatment
* History of recent temporal ischemic attack or malignant diseases (< 5 yrs)
* Celiac disease, or allergy or intolerance to the ingredients of the test products
* Medically prescribed diet/medication for slimming or a special diet like very low calorie diet or obesity drug, or vegan and gluten-free diet
* Subjects with alcohol abuse (> 4 portion per day)
* Pregnancy or planned pregnancy or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percentage change in serum LDL cholesterol | 4 weeks

SECONDARY OUTCOMES:
Absolute change in serum LDL cholesterol (mmol/l) | 4 weeks
Absolute and percentage change in serum total, HDL- and non-HDL cholesterol and serum total triglycerides | 4 weeks

REFERENCES:
- [Derived] Sarkkinen E, Lyyra M, Nieminen S, Kuusisto P, Wester I. Cereal-Based Snack Bar with Added Plant Stanol Ester (Benecol(R)) Consumed between Meals Lowers Serum Total and LDL Cholesterol Effectively in Mildly to Moderately Hypercholesterolemic Subjects. Cholesterol. 2018 May 2;2018:1463628. doi: 10.1155/2018/1463628. eCollection 2018. PMID 29854447